CLINICAL TRIAL: NCT00682292
Title: Multicenter Randomized Study to Compare Induction Therapy With Polyclonal Antithymocytes Globulins (ATG) Versus Monoclonal Anti-IL2R Antibody (Daclizumab) in a Triple Drug Regimen in Renal Transplant Recipients With High Immunological Risk.
Brief Title: Daclizumab Versus Thymoglobulin in Renal Transplant Recipients With High Immunological Risk
Acronym: TAXI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Erasme University Hospital (Other)
Responsible Party: Noël Christian, MD, PhD, Professor of Nephrology, University Hospital of Lille
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHLillle; CRG020600038
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2004-02

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation; Immunisation; Acute rejection; Induction therapy; Thymoglobulin; Daclizumab; Rejection in sensitized renal transplant recipients
MeSH Terms: interventions — thymoglobulin; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, ATG (Active Comparator): Thymoglobulin induction during 8 days (1.25 mg/kg per day) associated with tacrolimus, mycophenolate mofetil and steroids
  Interventions: Drug: Thymoglobulin (ATG)
- 2, Daclizumab (Active Comparator): Dacluzamb induction (five infusions, 1 mg/kg per infusion) associated with tacrolimus, mycophenolate mofetil and steroids
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Thymoglobulin (ATG) — Thymoglobulin: 1.25 mg/kg per day from day 0 to day 7 post transplantation
  Other Names: Thymoglobulin, Genzyme
  Arms: 1, ATG
Drug: Daclizumab — Daclizumab: 1mg/kg at day 0, 14, 28, 42 and 56 post transplantation
  Other Names: Zenapax, Roche
  Arms: 2, Daclizumab

SUMMARY:
To compare renal allograft rejection rates during the first year among high-immunological risk recipients between patients who received either ATG or the anti-IL2R mAb daclizumab.

DETAILED DESCRIPTION:
The objective of this randomized, multi-center trial is to directly compare the ATG, Thymoglobulin, with the anti-CD25 mAb, daclizumab, in a high-risk, HLA-sensitized renal transplant population, in order to elucidate whether there is any significant difference in the incidence of acute rejection after one year.

Eligible patients were randomized (1:1) to receive either ATG (1.25 mg/kg/d from day 0 to day 7) or daclizumab (1 mg/kg at days 0, 14, 28, 42 and 56). Maintenance immunosuppression comprised tacrolimus, MMF and prednisone. The study's primary endpoint was the incidence of biopsy-proven acute rejection at one year.

ELIGIBILITY:
Inclusion Criteria:

1. Third or fourth renal graft or
2. Current anti-HLA antibodies above or equal to 30% at the last evaluation or
3. Peak anti-HLA antibodies above or equal to 50% at the last evaluation or
4. A second graft if the first was lost within 2 years because of rejection.
5. Patients who gave their informed consent and are able to understand the scope of the study

Exclusion Criteria:

1. Transplantation from living donors or recipients of multiple grafts or patients who already have received another (non-renal) allograft.
2. Transplantation from a non-heart beating donor
3. Transplantation of two kidneys from the same donor
4. Patients with generalized infection at the time of transplantation
5. Women in child-bearing age who do not plan to use efficient contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2001-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-proven acute allograft rejection during the first post-transplant year | acute rejection proved by graft biopsy

SECONDARY OUTCOMES:
Proportion of patients who experienced an acute rejection episode, whether confirmed by biopsy or not at 1 year. | graft dysfunction
Proportion of patients who experienced more than one episode of acute allograft rejection | graft dysfunction, biopsies
Proportion of patients who experienced an acute rejection episode that required therapy by anti-lymphocyte antibodies (ATG or OKT3) | number of anti-lymphocyte treatment required for acute rejection episodes
Number of acute rejection episodes per therapeutic arms and mean number of acute rejection episode per patient in each arm | graft dysfunction and biopsies
Banff grade of the first rejection episode | graft biopsy
Incidence of adverse events in the two treatment arms at 1 year | number of adverse events reported by the investigators
Incidence of delayed graft function | number of patient who required hemodialysis during the first week post transplantation
Graft function at 1 year | serum creatinine and estimated glomerular filtration rate
Graft and patient survival at 1 year | number of graft failures and/or deaths

CONTACTS AND LOCATIONS:
Overall Officials: Christian Noël, MD, PhD, Principal Investigator — University Hospital of Lille, France; Daniel Abramowicz, MD, PhD, Principal Investigator — Erasme Hospital, Bruxelles, Belgium
Locations (1):
- University Hospital of Lille, Lille, France